CLINICAL TRIAL: NCT01374685
Title: Family Communication of Hereditary Cancer Risk Among African Americans
Brief Title: Family Communication of Hereditary Breast and Ovarian Cancer Risk Among African Americans
Status: Terminated | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911186; 11-HG-N186
Record Dates: First submitted 2011-06-15; First posted 2011-06-16 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2016-01-07

CONDITIONS: Ovarian Neoplasm; Cancer Genetics; Breast Cancer
Keywords: BRCA1; BRCA2; Breast Cancer; African American; Women
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

- Certain genetic mutations are linked to higher rates of cancer. It is important for people with these mutations to tell their families about it. This is because others in the family may also be at greater risk for developing these cancers. They can also pass these genes to their own children. But not much is known about how African Americans tell their family members about the results of their genetic testing. The information from this study can be used to improve genetic counseling services. These services will then be more effective in early cancer detection and prevention in the African American community.

Objectives:

- To learn more about how African Americans who have tested positive for BRCA1/2 mutations tell their families about their genetic risk.

Eligibility:

- African American (or of African descent) women who recently received positive test results for BRCA1/2 mutations.

Design:

* Participants will be screened with a basic medical history.
* They will be asked general questions about their personal and family history. These include questions on marital and health insurance status, education, and income.
* Those in the study will have a 45- to 60-minute phone interview. They will answer questions about how they told their family members about their genetic test results. They will also be asked what that experience was like.

DETAILED DESCRIPTION:
The ways in which family members communicate with one another about hereditary cancer risk may have a significant impact on screening use and choices about predictive genetic testing. There have been many studies examining aspects of family communication of hereditary cancer risk but few have included a significant number of African American families. The lack of studies addressing how African American patients communicate about genetic risks for cancer with their relatives is a hindrance to facilitating communication strategies in this patient population. The proposed study is a mixed methods investigation aimed at understanding how communication of hereditary breast and ovarian cancer risk occurs in African American families. This study will seek to describe how African American women communicate with their family members about the information received during the genetic counseling process for BRCA1/2 genetic testing by analyzing data from two sources. The data collected from data source one of this study will be from female analogue clients who were recruited from the general population in Baltimore, Maryland to watch a videotape of a pre-test cancer genetic counseling session. The analogue clients were asked to imagine they were the patients in the visit and to respond to several open-ended questions about what they would tell their family members about what they learned from the session. A quantitative content analysis of the data from the open-ended responses will be conducted to identify the frequency of commonly stated words, phrases and concepts related to the respondents characterization of the content of their family communication. From data source one of this study, we will obtain information on what women report they would share with their family members and the words they report they would use. Data source two of this study will involve in-depth qualitative interviews with 40 African American women who have tested positive for a BRCA1/2 mutation. These interviews will seek to understand how test results and information from the genetic counseling process were actually shared with family members. These interviews will seek to not only further describe what information individuals reported sharing with their family members but also how the process of communication unfolded. From these two forms of data, this study will describe the family communication process of hereditary cancer risk among African American women.

ELIGIBILITY:
* INCLUSION CRITERIA:

Understands and speaks English

African American

Women

18 years or older

Has had genetic testing for BRCA1/2 mutations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-06-07; Study Completion 2016-01-07

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B Biesecker, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Antoniou A, Pharoah PD, Narod S, Risch HA, Eyfjord JE, Hopper JL, Loman N, Olsson H, Johannsson O, Borg A, Pasini B, Radice P, Manoukian S, Eccles DM, Tang N, Olah E, Anton-Culver H, Warner E, Lubinski J, Gronwald J, Gorski B, Tulinius H, Thorlacius S, Eerola H, Nevanlinna H, Syrjakoski K, Kallioniemi OP, Thompson D, Evans C, Peto J, Lalloo F, Evans DG, Easton DF. Average risks of breast and ovarian cancer associated with BRCA1 or BRCA2 mutations detected in case Series unselected for family history: a combined analysis of 22 studies. Am J Hum Genet. 2003 May;72(5):1117-30. doi: 10.1086/375033. Epub 2003 Apr 3. PMID 12677558
- [Background] Armstrong K, Micco E, Carney A, Stopfer J, Putt M. Racial differences in the use of BRCA1/2 testing among women with a family history of breast or ovarian cancer. JAMA. 2005 Apr 13;293(14):1729-36. doi: 10.1001/jama.293.14.1729. PMID 15827311
- [Background] Barnes J, Kroll L, Burke O, Lee J, Jones A, Stein A. Qualitative interview study of communication between parents and children about maternal breast cancer. BMJ. 2000 Aug 19-26;321(7259):479-82. doi: 10.1136/bmj.321.7259.479. PMID 10948027